CLINICAL TRIAL: NCT01137396
Title: Modafinil, Sleep Architecture and Cocaine Relapse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0911005989; DA011744-08
Record Dates: First submitted 2010-06-03; First posted 2010-06-04 (Estimated); Results first posted 2016-04-27 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-03

CONDITIONS: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Modafinil; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Modafinil (Experimental)
  Interventions: Drug: Modafinil; Behavioral: Cognitive Behavioral Therapy
- Placebo (Placebo Comparator)
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Drug: Modafinil — Modafinil 400mg PO QDaily following up-titration for ~8weeks
  Arms: Modafinil
Behavioral: Cognitive Behavioral Therapy — Once weekly cognitive behavioral therapy for cocaine dependence

SUMMARY:
The medication modafinil has been shown to reduce cocaine use in some cocaine users. The investigators have shown that modafinil taken in the morning improves sleep in chronic cocaine users. The investigators hypothesize that the beneficial effects of modafinil in reducing cocaine use may be related to specific effects modafinil has on sleep. This study will measure sleep and cocaine use in cocaine dependent persons who are trying to stop using cocaine, and will test the connection between modafinil's effects on sleep and cocaine use.

ELIGIBILITY:
Inclusion Criteria:

* 25-50 years of age;
* voluntary, written, informed consent;
* seeking but not currently enrolled in treatment for cocaine use;
* self-reported, current use of cocaine by smoked or intravenous route at least one time each week in the past month, with ≥1g used within a single 24-hour period and ≥3g used in the month;
* positive urine test for cocaine (benzoylecognine) at the time of screening and study start
* dependence on cocaine in the past year as measured by a score ≥ 3 on the Severity of Dependence Scale(Kaye and Darke, 2002);
* chronic use in the past year as determined by self-reported use in at least 9 of the past 12 months;
* lifetime diagnosis of cocaine dependence with a duration of at least 2 years as determined by the Structured Clinical Interview for DSM-IV (SCID).

Exclusion Criteria:

* evidence of any neurological condition or a chronic medical condition including diabetes, cardiovascular disease or history of cardiac problems, HIV-seropositivity, liver disease, hypertension, asthma requiring daily medication, dementia, movement disorder, history of head trauma with loss of consciousness, sleep apnea, narcolepsy, restless leg syndrome, periodic limb movement disorder, REM sleep disorder, pharmacological treatment for insomnia of any type within the past 6 months, glaucoma, severe respiratory insufficiency, seizure disorder, or if in the past three months they have taken any medications that affect sleep, or are currently taking any regularly dosed prescription medication or any prn medication that is used on average more than 1x/week
* evidence of chronic sleep disorder including sleep apnea, narcolepsy, periodic limb movement disorder, restless leg syndrome as determined by medical history, Sleep Disorders Questionnaire(Douglass, 1994), or by polysomnography (following enrollment)
* current dependence on any drugs other than cocaine or nicotine or lifetime dependence on alcohol, benzodiazepines, or opiates, or any non-substance related Axis I disorder as determined by SCID
* current use of alcohol in excess of 3x/week AND 21 standard drinks/week in the past month or non-zero breathalyzer at screening or study start
* current use of cannabis in the past month
* positive urine toxicology test for opiates, methadone, amphetamines, barbiturates, benzodiazepines, PCP, methaquolone, and propoxyphene at the time of screening or positive test for any of those listed plus cannabis at the time of study start
* pregnancy as determined by serum β-HCG at screening or lactating per report
* females: unwillingness to use barrier contraceptives during sexual intercourse for the duration of the study
* known hypersensitivity to modafinil.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2010-04; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Morgan, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Angarita GA, Canavan SV, Forselius E, Bessette A, Pittman B, Morgan PT. Abstinence-related changes in sleep during treatment for cocaine dependence. Drug Alcohol Depend. 2014 Jan 1;134:343-347. doi: 10.1016/j.drugalcdep.2013.11.007. Epub 2013 Nov 17. PMID 24315572

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo: Placebo medication Qdaily for ~8weeks
  Cognitive Behavioral Therapy: Once weekly cognitive behavioral therapy for cocaine dependence
Period: Overall Study
Arm/Group | Modafinil | Placebo
Started | 30 | 27
Completed | 22 | 25
Not Completed | 8 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Modafinil | Placebo | Total
Number analyzed (Participants) | 30 | 27 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (7) | 44 (7) | 43 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 23 | 21 | 44

OUTCOME MEASURES:

1. Primary Outcome: %Cocaine Free Urines
Time Frame: 3x/week
Measure: Mean (Standard Error); unit: percent
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 22 | 25
percent | 52 (9) | 26 (7)

2. Secondary Outcome: Change in N3 (Slow-wave) Sleep Time
Time Frame: change from week 1 to week 2 of inpatient treatment
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 22 | 25
minutes | 16 (4) | -2.5 (4)

ADVERSE EVENTS:
Arm/Group | Modafinil | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/27
Other Adverse Events (participants affected / at risk) | 0/30 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No